CLINICAL TRIAL: NCT03838731
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study in Cat-Allergic Patients With Asthma to Evaluate the Efficacy of a Single Dose of REGN1908-1909 to Reduce Bronchoconstriction Upon Cat Allergen Challenge
Brief Title: Study in Cat-Allergic Patients With Asthma to Evaluate the Efficacy of a Single Dose of REGN1908-1909 to Reduce Bronchoconstriction Upon Cat Allergen Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1908-1909-ALG-1703; 2018-002477-22 (EudraCT Number)
Record Dates: First submitted 2019-02-09; First posted 2019-02-12 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Cat Allergy; Mild Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- REGN1908-1909 (Experimental)
  Interventions: Drug: REGN1908-1909
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN1908-1909 — Single subcutaneous (SC) dose of REGN1908 and REGN1909
  Arms: REGN1908-1909
Drug: Placebo — Single subcutaneous (SC) dose of matching placebo
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the prophylactic efficacy of REGN1908-1909 (anti-Fel d 1) administered as a single dose on day 1 in cat-allergic asthmatic patients not living with a cat in the prevention of a Controlled Cat Allergen Challenge-induced early asthmatic response (EAR) assessed by measures of lung function (FEV1) compared to placebo-treated patients.

Secondary Efficacy Objectives:

* To evaluate the prophylactic efficacy of REGN1908-1909 administered as a single dose on day 1 in cat-allergic asthmatic patients not living with a cat, in the prevention of a Controlled Cat Allergen Challenge-induced: Allergic rhinitis and Ocular symptoms
* To evaluate the prophylactic efficacy of REGN1908-1909 administered as a single dose on day 1 in cat-allergic asthmatic patients not living with a cat to increase the exposure to cat allergen, measured as a product of minute ventilation and time, required to induce EAR in a Controlled Cat Allergen Challenge as compared to placebo patients

Secondary Safety Objective:

* To evaluate the safety and tolerability of REGN1908-1909 vs. placebo in patients with cat allergen-triggered asthma

ELIGIBILITY:
Key Inclusion Criteria:

* Documented or patient reported history (for at least 2 years) of symptomatic cat allergen-triggered asthma with rhinitis with or without conjunctivitis
* No cat exposure at home for the past year and must continue having no exposure at home during the study; cat exposure outside of the home shall be avoided for at least one week prior to any Cat Allergen Challenge and during the defined follow-up period
* Less than 10 pack-years of smoking history

Key Exclusion Criteria:

* Positive human immunodeficiency virus (HIV) test
* Positive hepatitis test (HBsAg and hepatitis C antibody)
* History of significant multiple and/or severe allergies (including latex gloves) or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food
* Participation in a prior REGN1908-1909 clinical trial
* History of severe anaphylactic or severe asthmatic reactions to cat exposure
* Active lung disease other than asthma
* Treatment with an investigational drug within 2 months or within 5 half-lives (if known), whichever is longer, prior to screening
* Persistent chronic or recurring acute infection requiring treatment with antibiotics, antivirals, or antifungals, or any untreated respiratory infections within 4 weeks prior to screening
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest, and/or hypoxic seizures
* Treatment of asthma requiring systemic (oral or parenteral) corticosteroid treatment more than twice within 12 months or once within 3 months prior to screening or has been hospitalized or has attended the ER/Urgent Care facility for asthma more than twice in prior 12 months before screening.
* History of hypersensitivity to corticosteroids or antihistamines, or drug treatment excipient

Note: Other protocol defined Inclusion/Exclusion Criteria Apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Site, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual de-identified participant data will be made available once the indication has been approved by a regulatory body, if there is participant consent and there is not a reasonable likelihood of participant re-identification
Access Criteria: Qualified researchers may request access to study documents (including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan) that support the methods and findings reported in a manuscript. Individual de-identified participant data will be made available once the indication has been approved by a regulatory body, if there is participant consent and there is not a reasonable likelihood of participant re-identification
URL: https://vivli.org/

REFERENCES:
- [Derived] de Blay FJ, Gherasim A, Domis N, Meier P, Shawki F, Wang CQ, Orengo JM, DeVeaux M, Ramesh D, Jalbert JJ, Kamal MA, Abdallah H, Dingman R, Perlee L, Weinreich DM, Herman G, Yancopoulos GD, O'Brien MP. REGN1908/1909 prevented cat allergen-induced early asthmatic responses in an environmental exposure unit. J Allergy Clin Immunol. 2022 Dec;150(6):1437-1446. doi: 10.1016/j.jaci.2022.06.025. Epub 2022 Aug 4. PMID 35934082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 130 participants were screened for study eligibility. Screen failures were mostly attributed to eligibility criteria not being met. The study was conducted at one site in France.
Pre-assignment Details: A total of 56 participants were randomized in a 1:1 ratio to receive a single dose of either 600 milligrams (mg) of REGN1908-1909 or matching placebo.
Groups:
- Placebo: Participants received a single dose of matching placebo
- REGN1908-1909 600 mg: Participants received a single 600 mg dose of REGN1908-1909
Period: Overall Study
Arm/Group | Placebo | REGN1908-1909 600 mg
Started | 27 | 29
Completed | 26 | 28
Not Completed | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal of consent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | REGN1908-1909 600 mg | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.2 (8.8) | 28.4 (7.1) | 29.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 24 | 27 | 51
  Other | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Early Asthmatic Response (EAR) Upon Controlled Cat Allergen Challenge in an Environmental Exposure Unit (EEU) on Day 8
Description: Time to EAR was defined as the time to a ≥20% reduction in FEV1 or when the participant voluntarily departed the EEU due to clinically significant allergic and/or asthmatic symptoms.
Time Frame: Day 8
Population: Full analysis set: included all randomized participants who received any investigational product and had completed the Day 8 Cat Allergen Challenge.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | REGN1908-1909 600 mg
Number analyzed (Participants) | 27 | 29
Minutes | 51 [33.92 to 70.70] | NA [130.87 to NA] — The median time to EAR could not be estimated in the REGN1908-1909 arm at the day 8 visit since a majority of participants were able to tolerate the full 4 hours of cat allergen exposure, the maximum time allowed in the EEU per protocol, without experiencing an EAR (censored at 4 hours)
Statistical Analysis 1: Comparison: Placebo vs REGN1908-1909 600 mg; Test type: Superiority; p = 0.0083, Cox Proportional Hazard; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.17 to 0.77]

2. Secondary Outcome: Time to EAR Upon Controlled Cat Allergen Challenge in an EEU on Days 29, 57, and 85
Description: as for outcome 1
Time Frame: Days 29, 57 and 85
Population: Full analysis set: included all randomized participants who received any investigational product and had completed the Day 8 Cat Allergen Challenge. Here "n" = number of evaluable participants analyzed at each time point
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | REGN1908-1909 600 mg
Number analyzed (Participants) | 27 | 29
Minutes
  Day 29: number analyzed (Participants) | 25 | 29
  Day 29 | 41 [31.38 to 61.13] | NA [131.22 to NA] — Time to EAR, post-baseline, was censored at 4 hours if the participant remained in the EEU for the maximum time and did not experience an EAR. Baseline EEU maximum exposure was 2 hours.
  Day 57: number analyzed (Participants) | 26 | 27
  Day 57 | 56 [40.52 to 80.63] | 232 [81.05 to NA] — Time to EAR, post-baseline, was censored at 4 hours if the participant remained in the EEU for the maximum time and did not experience an EAR. Baseline EEU maximum exposure was 2 hours.
  Day 85: number analyzed (Participants) | 24 | 26
  Day 85 | 41 [31.03 to 60.93] | NA [90.97 to NA] — Time to EAR, post-baseline, was censored at 4 hours if the participant remained in the EEU for the maximum time and did not experience an EAR. Baseline EEU maximum exposure was 2 hours.
Statistical Analysis 1: Comparison: Placebo vs REGN1908-1909 600 mg; Day 29; Test type: Superiority; p < 0.0001, Cox Hazard Model; Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.12 to 0.48]
Statistical Analysis 2: Comparison: Placebo vs REGN1908-1909 600 mg; Day 57; Test type: Superiority; p = 0.0222, Cox Hazard Model; Hazard Ratio (HR) = 0.45, 95% CI [0.22 to 0.89]
Statistical Analysis 3: Comparison: Placebo vs REGN1908-1909 600 mg; Day 85; Test type: Superiority; p = 0.0003, Cox Hazard Model; Hazard Ratio (HR) = 0.27, 95% CI [0.13 to 0.56]

3. Secondary Outcome: Percent Change in Normalized Area Under the Curve (AUC) of Forced Expiratory Volume in 1 Second (FEV1) Induced by a Controlled Cat Allergen Challenge Over Exposure Interval From Baseline to Controlled Cat Allergen Challenge on Days 8, 29, 57, and 85
Description: The AUC was analyzed by mixed-effect model repeated measures (MMRM) with the treatment, time, treatment-by-time interaction, and day of challenge as factors and baseline FEV1 AUC as a continuous covariate.
Time Frame: Days 8, 29, 57, and 85
Population: Full analysis set; Here 'n' = number of evaluable participants analyzed at each time point. For each participant at each controlled cat allergen challenge, AUC was calculated over the time period of 0 to 2 hours, with last observation carried forward used to impute values out to 2 hours if the patients remained in EEU for less than 2 hours. The AUCs were calculated using the trapezoidal rule and were normalized by dividing by the length of time (2 hours).
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo | REGN1908-1909 600 mg
Number analyzed (Participants) | 27 | 29
Percentage of change
  Day 8 | 1.59 (2.58) | 15.15 (2.50)
  Day 29: number analyzed (Participants) | 25 | 29
  Day 29 | 0.46 (3.60) | 16.67 (3.43)
  Day 57: number analyzed (Participants) | 26 | 28
  Day 57 | 1.77 (3.55) | 14.07 (3.43)
  Day 85: number analyzed (Participants) | 24 | 26
  Day 85 | 0.20 (3.28) | 12.73 (3.14)
Statistical Analysis 1: Comparison: Placebo vs REGN1908-1909 600 mg; Test type: Superiority — Day 8; p < 0.001, MMRM; LS Mean Difference = 13.56, 95% CI 2-sided [6.35 to 20.77], Standard Error of Mean 3.59
Statistical Analysis 2: Comparison: Placebo vs REGN1908-1909 600 mg; Test type: Superiority — Day 29; p = 0.002, MMRM; LS Mean Difference = 16.21, 95% CI 2-sided [6.18 to 26.24], Standard Error of Mean 4.97
Statistical Analysis 3: Comparison: Placebo vs REGN1908-1909 600 mg; Test type: Superiority — Day 57; p = 0.016, MMRM; LS Mean Difference = 12.30, 95% CI 2-sided [2.40 to 22.20], Standard Error of Mean 4.94
Statistical Analysis 4: Comparison: Placebo vs REGN1908-1909 600 mg; Test type: Superiority — Day 85; p = 0.008, MMRM; LS Mean Difference = 12.54, 95% CI 2-sided [3.43 to 21.65], Standard Error of Mean 4.54

4. Secondary Outcome: Change in Normalized Area Under the Curve (AUC) of Forced Expiratory Volume in 1 Second (FEV1) Induced by a Controlled Cat Allergen Challenge Over Exposure Interval From Baseline to Controlled Cat Allergen Challenge on Days 8, 29, 57, and 85
Description: as for outcome 3
Time Frame: Days 8, 29, 57, and 85
Population: Full analysis set; Here "n" = number of evaluable participants analyzed at each time point. For each participant at each controlled cat allergen challenge, AUC was calculated over the time period of 0 to 2 hours, with last observation carried forward used to impute values out to 2 hours if the patients remained in EEU for less than 2 hours. The AUCs were calculated using the trapezoidal rule and were normalized by dividing by the length of time (2 hours).
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | Placebo | REGN1908-1909 600 mg
Number analyzed (Participants) | 27 | 29
Liters (L)
  Day 8 | 0.01 (0.06) | 0.38 (0.06)
  Day 29: number analyzed (Participants) | 25 | 29
  Day 29 | -0.03 (0.08) | 0.43 (0.08)
  Day 57: number analyzed (Participants) | 26 | 28
  Day 57 | 0.00 (0.08) | 0.34 (0.07)
  Day 85: number analyzed (Participants) | 24 | 26
  Day 85 | -0.05 (0.08) | 0.32 (0.08)
Statistical Analysis 1: Comparison: Placebo vs REGN1908-1909 600 mg; Day 8; Test type: Superiority; p < 0.001, MMRM; LS Mean Difference = 0.37, 95% CI 2-sided [0.21 to 0.53], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Placebo vs REGN1908-1909 600 mg; Day 29; Test type: Superiority; p < 0.001, MMRM; LS Mean Difference = 0.46, 95% CI 2-sided [0.23 to 0.68], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Placebo vs REGN1908-1909 600 mg; Day 57; Test type: Superiority; p = 0.002, MMRM; LS Mean Difference = 0.34, 95% CI 2-sided [0.13 to 0.55], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Placebo vs REGN1908-1909 600 mg; Day 85; Test type: Superiority; p = 0.002, MMRM; LS Mean Difference = 0.37, 95% CI 2-sided [0.15 to 0.47], Standard Error of Mean 0.11

5. Secondary Outcome: Change From Baseline in the Normalized AUC of Patient-Assessed Nasal Symptoms Induced by a Controlled Cat Allergen Challenge Over the Exposure Interval to the Controlled Cat Allergen Challenge on Days 8, 29, 57, and 85
Description: Individual nasal symptoms, including rhinorrhea, nasal congestion, nasal itching, and sneezing were evaluated on a 4-point Likert scale (0, none; 1, mild; 2, moderate; and 3, severe) and combined to give the Total Nasal Symptom Score (TNSS) with a maximum score of 12. Scale range is 0-12. The higher the score, the more severe the symptoms.
Time Frame: Days 8, 29, 57 and 85
Population: Full analysis set; Here 'n' = number of evaluable participants analyzed at each time point. For each participant at each controlled cat allergen challenge, AUC was calculated over the time period of 0 to 2 hours, with last observation carried forward used to impute values out to 2 hours if participants remained in EEU for less than 2 hours. AUCs were calculated using trapezoidal rule and were normalized by dividing by the length of time (2 hours).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | REGN1908-1909 600 mg
Number analyzed (Participants) | 27 | 29
Scores on a scale
  Day 8: number analyzed (Participants) | 25 | 26
  Day 8 | -0.71 (0.38) | -0.49 (0.38)
  Day 29: number analyzed (Participants) | 23 | 27
  Day 29 | -0.70 (0.37) | -1.39 (0.34)
  Day 57: number analyzed (Participants) | 24 | 26
  Day 57 | -0.93 (0.43) | -0.83 (0.43)
  Day 85: number analyzed (Participants) | 22 | 24
  Day 85 | -0.49 (0.43) | -1.37 (0.41)
Statistical Analysis 1: Comparison: Placebo vs REGN1908-1909 600 mg; Day 8; Test type: Superiority; p = 0.675, MMRM; LS Mean Difference = 0.22, 95% CI 2-sided [-0.85 to 1.29], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: Placebo vs REGN1908-1909 600 mg; Day 29; Test type: Superiority; p = 0.182, MMRM; LS Mean Difference = -0.68, 95% CI 2-sided [-1.70 to 0.33], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Placebo vs REGN1908-1909 600 mg; Day 57; Test type: Superiority; p = 0.866, MMRM; LS Mean Difference = 0.10, 95% CI 2-sided [-1.12 to 1.32], Standard Error of Mean 0.61
Statistical Analysis 4: Comparison: Placebo vs REGN1908-1909 600 mg; Day 85; Test type: Superiority; p = 0.146, MMRM; LS Mean Difference = -0.88, 95% CI 2-sided [-2.08 to 0.32], Standard Error of Mean 0.60

6. Secondary Outcome: Change From Baseline in the Normalized AUC in Patient-Assessed Ocular Symptoms Induced by a Controlled Cat Allergen Challenge Over the Exposure Interval to the Controlled Cat Allergen Challenge on Days 8, 29, 57, and 85
Description: Individual ocular symptoms for itching/burning, redness, swelling/puffiness, and tearing/watery eyes were evaluated on a 4-point Likert scale (0, none; 1, mild; 2, moderate; and 3, severe) and combined to give the TOSS, with a maximum score of 12. Score range is 0-12. The higher the score, the more severe the symptoms.
Time Frame: Days 8, 29, 57 and 85
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | REGN1908-1909 600 mg
Number analyzed (Participants) | 25 | 28
Scores on a scale
  Day 8: number analyzed (Participants) | 25 | 27
  Day 8 | -0.37 (0.17) | -0.23 (0.17)
  Day 29: number analyzed (Participants) | 23 | 28
  Day 29 | -0.43 (0.15) | -0.43 (0.14)
  Day 57: number analyzed (Participants) | 24 | 27
  Day 57 | -0.40 (0.15) | -0.34 (0.15)
  Day 85: number analyzed (Participants) | 22 | 25
  Day 85 | -0.36 (0.11) | -0.51 (0.10)
Statistical Analysis 1: Comparison: Placebo vs REGN1908-1909 600 mg; Day 8; Test type: Superiority; p = 0.572, MMRM; LS Mean Difference = 0.14, 95% CI 2-sided [-0.35 to 0.63], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs REGN1908-1909 600 mg; Day 29; Test type: Superiority; p = 0.997, MMRM; LS Mean Difference = -0.00, 95% CI 2-sided [-0.41 to 0.41], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Placebo vs REGN1908-1909 600 mg; Day 57; Test type: Superiority; p = 0.756, MMRM; LS Mean Difference = 0.07, 95% CI 2-sided [-0.36 to 0.49], Standard Error of Mean 0.21
Statistical Analysis 4: Comparison: Placebo vs REGN1908-1909 600 mg; Day 85; Test type: Superiority; p = 0.333, MMRM; LS Mean Difference = -0.15, 95% CI 2-sided [-0.46 to 0.16], Standard Error of Mean 0.15

7. Secondary Outcome: Mean Change From Baseline in Cat Allergen Quantity as Experienced by Participants During Exposure on Days 8, 29, 57, and 85
Description: Cat Allergen Exposure Tolerated in ng = Minute Ventilation (L/min) x Allergen Concentration (ng/m3) x Time in EEU (minutes), where 1 L/min = 0.001 m3/min. The change in cat allergen quantity (tolerated exposure) from the baseline Cat Allergen Challenge, will be analyzed using a similar MMRM model with treatment, visit and treatment by-visit interaction as factors and the cat allergen quantity tolerated in the baseline Controlled Cat Allergen Challenge as a covariate.
Time Frame: Days 8, 29, 57 and 85
Population: Full analysis set: included all randomized participants who received any investigational product and had completed the Day 8 Cat Allergen Challenge; Here "n" = number of evaluable participants analyzed at each time point
Measure: Least Squares Mean (Standard Error); unit: Nanograms (ng)
Arm/Group | Placebo | REGN1908-1909 600 mg
Number analyzed (Participants) | 27 | 29
Nanograms (ng)
  Day 8: number analyzed (Participants) | 24 | 24
  Day 8 | 19.55 (8.93) | 59.05 (8.70)
  Day 29: number analyzed (Participants) | 25 | 29
  Day 29 | 14.14 (8.67) | 68.21 (8.21)
  Day 57: number analyzed (Participants) | 26 | 26
  Day 57 | 21.94 (10.23) | 55.38 (9.93)
  Day 85: number analyzed (Participants) | 24 | 26
  Day 85 | 12.93 (9.29) | 54.03 (8.94)
Statistical Analysis 1: Comparison: Placebo vs REGN1908-1909 600 mg; Day 8; Test type: Superiority; p = 0.003, MMRM; LS Mean Difference = 39.50, 95% CI 2-sided [14.36 to 64.65], Standard Error of Mean 12.50
Statistical Analysis 2: Comparison: Placebo vs REGN1908-1909 600 mg; Day 29; Test type: Superiority; p < 0.001, MMRM; LS Mean Difference = 54.07, 95% CI 2-sided [30.01 to 78.12], Standard Error of Mean 11.97
Statistical Analysis 3: Comparison: Placebo vs REGN1908-1909 600 mg; Day 57; Test type: Superiority; p = 0.023, MMRM; LS Mean Difference = 33.44, 95% CI 2-sided [4.79 to 62.08], Standard Error of Mean 14.28
Statistical Analysis 4: Comparison: Placebo vs REGN1908-1909 600 mg; Day 85; Test type: Superiority; p = 0.003, MMRM; LS Mean Difference = 41.10, 95% CI 2-sided [15.10 to 67.09], Standard Error of Mean 12.92

8. Secondary Outcome: Percent Change in Cat Allergen Quantity as Experienced by Participants During Exposure on Days 8, 29, 57, and 85
Description: as for outcome 7
Time Frame: Days 8, 29, 57 and 85
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | Placebo | REGN1908-1909 600 mg
Number analyzed (Participants) | 27 | 29
Percentage of change
  Day 8: number analyzed (Participants) | 24 | 24
  Day 8 | 119.86 (73.22) | 325.29 (70.79)
  Day 29: number analyzed (Participants) | 25 | 29
  Day 29 | 93.62 (71.48) | 338.22 (68.26)
  Day 57: number analyzed (Participants) | 26 | 26
  Day 57 | 118.08 (69.58) | 301.11 (67.11)
  Day 85: number analyzed (Participants) | 24 | 26
  Day 85 | 76.75 (82.08) | 317.76 (78.84)
Statistical Analysis 1: Comparison: Placebo vs REGN1908-1909 600 mg; Day 8; Test type: Superiority; p = 0.049, MMRM; LS Mean Difference = 205.43, 95% CI 2-sided [0.69 to 410.17], Standard Error of Mean 102.09
Statistical Analysis 2: Comparison: Placebo vs REGN1908-1909 600 mg; Day 29; Test type: Superiority; p = 0.017, MMRM; LS Mean Difference = 244.60, 95% CI 2-sided [45.60 to 443.59], Standard Error of Mean 99.05
Statistical Analysis 3: Comparison: Placebo vs REGN1908-1909 600 mg; Day 57; Test type: Superiority; p = 0.064, MMRM; LS Mean Difference = 183.03, 95% CI 2-sided [-11.29 to 377.35], Standard Error of Mean 96.91
Statistical Analysis 4: Comparison: Placebo vs REGN1908-1909 600 mg; Day 85; Test type: Superiority; p = 0.039, MMRM; LS Mean Difference = 241.01, 95% CI 2-sided [12.44 to 469.57], Standard Error of Mean 114.00

9. Secondary Outcome: Number of Non-Serious and Serious Treatment-Emergent Adverse Events (TEAEs) Through End of Study
Description: Adverse events and serious adverse events were collected from the time of informed consent signature and then at each visit until the end of the study with the exception of symptoms that occurred in response to the EEU within 24 hours following the EEU.
Time Frame: Baseline to 16 weeks
Population: Safety Analysis Set (SAF): included all participants who received any investigational product and were analyzed as treated.
Measure: Number; unit: Events
Arm/Group | Placebo | REGN1908-1909 600 mg
Number analyzed (Participants) | 27 | 29
Events
  Non-serious TEAEs | 66 | 76
  Serious TEAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (day 1) to the end of study (week 16)
Groups:
- REGN1908-1909 600mg: Participants received a single 600 mg dose of REGN1908-1909
Arm/Group | Placebo | REGN1908-1909 600mg
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 19/27 | 22/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | REGN1908-1909 600mg (N=29)
Asthma (Respiratory, thoracic and mediastinal disorders) | 16 (35) | 11 (19)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Influenza like illness (General disorders) | 4 (4) | 3 (3)
Injection site pain (General disorders) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 5 (5)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03838731/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT03838731/SAP_001.pdf